CLINICAL TRIAL: NCT01406262
Title: A Randomized, Double-blind, Parallel, Nested Crossover Study to Investigate the Effect of Albiglutide on Cardiac Repolarization (Corrected QT Interval) Compared With Placebo in Healthy Male and Female Subjects: A Thorough ECG Study Employing Placebo, Albiglutide, and a Positive Control (Moxifloxacin)
Brief Title: Albiglutide Thorough ECG Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 107085
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: albiglutide; QT interval; cardiac repolarization; ECG study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albiglutide + moxifloxacin placebo (Active Comparator): Once weekly subcutaneous injection of albiglutide for 6 weeks plus oral tablet of moxifloxacin matching placebo on Days -1 and 40
  Interventions: Biological: Albiglutide
- Albiglutide matching placebo + moxifloxacin (Active Comparator): Once weekly subcutaneous injection of albiglutide matching placebo for 6 weeks, given with oral 400mg moxifloxacin tablet on Day -1 and moxifloxacin matching placebo on Day 40, or weekly albiglutide matching placebo for 6 weeks plus oral moxifloxacin matching placebo on Day -1 then oral 400mg moxifloxacin on Day 40
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Biological: Albiglutide — once weekly subcutaneous injection
  Arms: Albiglutide + moxifloxacin placebo
Drug: Moxifloxacin — oral tablet
  Arms: Albiglutide matching placebo + moxifloxacin

SUMMARY:
This study is designed to investigate the effect of treatment with albiglutide on the cardiac repolarization (corrected QT interval) in healthy male and female subjects. Moxifloxacin, a positive control, or moxifloxacin placebo will be given in order to validate the ability of the study to detect a change in the corrected QT interval.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind study designed to investigate the effect of treatment with albiglutide given weekly over 6 weeks on the cardiac repolarization (corrected QT interval) in healthy male and female subjects. Moxifloxacin, a positive control, or moxifloxacin placebo will be given in order to validate the ability of the study to detect a change in the corrected QT interval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or nonpregnant, nonlactating female
* Subject considered to be in good health as judged by the absence of clinically significant diseases or clinically significant abnormal laboratory values
* BMI is ≥18 kg/m2 and ≤30 kg/m2
* Nonsmoker

Exclusion Criteria:

* Positive test results for hepatitis B, hepatitis C, or human immunodeficiency virus
* History of arrythmia or use of antiarrhythmic agents
* History of any anaphylactic reaction to any drug
* History of significant cardiovascular or pulmonary dysfunction
* Current or chronic history of liver disease , renal disease, CNS disorders, thyroid dysfunction, rheumatoid arthritis
* History of alcohol or substance abuse
* History of GI surgery that could influence gastric emptying
* Female and using oral contraception (combined or progestogen only), implants or levonorgestrel, or injectable progesterone, or hormone replacement therapy
* History of pancreatitis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2011-12-29 (Actual); Study Completion 2011-12-29 (Actual)

PRIMARY OUTCOMES:
QTc interval | 6 weeks
  Measurement of cardiac repolarization after albiglutide dosing

SECONDARY OUTCOMES:
QTc interval | Day 4
  Measurement of cardiac repolarization after albiglutide dosing
QT interval | Day -1 and Day 40
  Determination of the effect of moxifloxacin on cardiac repolarization
Number of participants with adverse events | 6 weeks
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Results for study 107085 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/107085?search=study&study_ids=107085#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 107085 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107085 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107085 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107085 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107085 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107085 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107085 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register